CLINICAL TRIAL: NCT04785300
Title: ALSENLITE: An Open-Label Pilot Study of Senolytics for Alzheimer's Disease
Brief Title: ALSENLITE: Senolytics for Alzheimer's Disease
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Vijay K. Ramanan, Assistant Professor of Neurology, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-003394
Record Dates: First submitted 2021-03-04; First posted 2021-03-05 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Mild Cognitive Impairment; Alzheimer Disease
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease | interventions — Dasatinib; Quercetin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dasatinib plus Quercetin Treatment Goup (Experimental): Subjects with MCI or Alzheimer's disease will take Dasatinib and Quercetin by mouth at the same times for 2 days out of every 15 days for 6 cycles lasting for a total of 77 days (12 concurrent doses of each agent).
  Interventions: Drug: Dasatinib; Drug: Quercetin

INTERVENTIONS:
Drug: Dasatinib — 100 mg capsule daily for 2 consecutive days administered orally every 15 days (2 days on drug, 13 days off) for 6 cycles
Drug: Quercetin — Four 250 capsules once daily (total daily dosage 1000 mg) administered orally for 2 consecutive days every 15 days (2 days on drug, 13 days off) for 6 cycles

SUMMARY:
This study is being done to evaluate the safety and feasibility of using Dasatinib and Quercetin together in subjects with Mild Cognitive Impairment (MCI) or Alzheimer's disease.

DETAILED DESCRIPTION:
The underlying processes driving chronic neurodegeneration in Alzheimer's disease (AD) and related neurodegenerative disorders are largely unknown. Aging is the major risk factor for AD. Moreover, individuals with AD suffer from significantly more co-morbid conditions than demographically matched older adults. This study is an open-label pilot study of intermittent administration of the senolytic drug regimen Dasatinib (D) + Quercetin (Q) in symptomatic adults over 55 with clinical diagnosis of probable Alzheimer's Disease and Alzheimer's biomarker positivity by tau-PET.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women of age 55 years and older at the time of enrollment
2. Clinical diagnosis of symptomatic probable AD (MMSE 26 to 15 or Short Test of Mental Status 31 to 15 inclusive and/or Clinical Dementia Rating Scale/CDR = 0.5 to 2, inclusive)
3. Not on cholinesterase inhibitors or memantine; or if on cholinesterase inhibitors and/or memantine, on a stable dose for at least three months
4. Body Mass Index (BMI) within range of 19 - 50 kg/ m2
5. Participants must be accompanied by a LAR designated to sign informed consent and to provide study partner reported outcomes at all visits
6. Participants must have no plans to travel over the ~3 months between Visits 3 and 14 that interfere with study visits
7. Tau positivity by brain PET imaging
8. Adequate blood counts i.e. platelets > 50,000 per microliter; HB > 9/dL, and ANC > 1000 per microliter
9. Availability and consent from a LAR.

Exclusion Criteria:

1. Unwilling or unable to give informed consent
2. Pregnancy
3. QTc > 450 msec on baseline ECG
4. MRI contraindications
5. Presence of uncontrolled psychiatric disorder (as per clinical judgment)
6. Presence of uncontrolled systemic lupus erythematosus (as per clinical judgment)
7. Substance or alcohol abuse (current alcohol use > 3 alcoholic beverage/day or > 21 per week and as per clinical judgment)
8. Hearing, vision, or motor deficits despite corrective devices (as per clinical judgment)
9. Myocardial infarction, angina, stroke, or transient ischemic attack in the past 6 months
10. Chronic heart failure (as per clinical judgment)
11. Neurologic, musculoskeletal, or other condition that limits subject's ability to complete study physical assessments (as per clinical judgment)
12. Positive SARS-CoV-2 test within 30 days prior to enrollment
13. AST/ALT > 2.5x upper limit normal
14. Presence of significant liver disease with total bilirubin > 2X upper limit or as per clinical judgment
15. Inability to tolerate oral medication (as per clinical judgment)
16. Abnormality in any of the screening laboratory studies (see section 6.21.2) or as per clinical judgment
17. Malabsorption (as per clinical judgment)
18. Known human immunodeficiency virus infection (as per clinical judgment)
19. Known active hepatitis B or C infection
20. Invasive fungal or viral infection (as per clinical judgment)
21. Known hypersensitivity or allergy to D or Q
22. Uncontrolled pleural/pericardial effusions or ascites (as per clinical judgment)
23. New/active invasive cancer except non-melanoma skin cancers
24. Inability to tolerate oral medications (as per clinical judgment)
25. Currently taking AND unable to safely hold any of the medications listed in Appendix 1 during the days IP is administered and for 36 hours after IP administration.
26. Uncontrolled diabetes (defined as HbA1c > 7% or as per clinical judgment).
27. Gastric bypass/reduction
28. Crohn's disease
29. Myopathies (increased or low calcium, vitamin D deficiency, elevated creatine kinase or ESR) (as per clinical judgment)
30. eGFR < 10 ml/ min/ 1.73 m2
31. Creatinine clearance < 60 mL/min/1.73 m2
32. Subjects on therapeutic doses of anticoagulants (e.g., warfarin, heparin, low molecular weight heparin, factor Xa inhibitors, etc.)
33. On antiplatelet agents (e.g., full dose Aspirin, Clopidogrel etc.). Baby aspirin (81 mg), if absolutely necessary from cardiac perspective, will be allowed
34. Presence of any condition that the Investigator believes would put the subject at risk or would preclude the patient from successfully completing all aspects of the trial

Involvement of special vulnerable populations: We will not involve special vulnerable populations, such as fetuses, neonates, pregnant women, children, prisoners, institutionalized individuals, or others who may be considered vulnerable populations except for patients with dementia. Therefore, availability and consent from a LAR is an inclusion criterion.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-07-06 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | 11 weeks
  Safety evaluations will be conducted including assessment for adverse events, compliance to the study drug regimen, physical examinations or assessments, vital signs, and laboratory assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Vijay K. Ramanan, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Andrews TD, Day GS, Irani SR, Kanekiyo T, Hickson LJ. Uremic Toxins, CKD, and Cognitive Dysfunction. J Am Soc Nephrol. 2025 Jun 1;36(6):1208-1226. doi: 10.1681/ASN.0000000675. Epub 2025 Feb 26. PMID 40009460
- [Derived] Guerrero A, De Strooper B, Arancibia-Carcamo IL. Cellular senescence at the crossroads of inflammation and Alzheimer's disease. Trends Neurosci. 2021 Sep;44(9):714-727. doi: 10.1016/j.tins.2021.06.007. Epub 2021 Aug 5. PMID 34366147